CLINICAL TRIAL: NCT04251520
Title: The Role of the Pharmacist and Pharmacogenomics in the Care of Seriously Ill Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark K. Edwin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-010761
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Palliative Medicine
Keywords: Pharmacogenomics; Symptom management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Standard care by Palliative Medicine physician
- Intervention Group A (Experimental): Standard care by Palliative medicine physician plus pharmacist review of medications
  Interventions: Other: Pharmacist review
- Intervention Group B (Experimental): Standard care by Palliative medicine plus pharmacogenomics testing and pharmacist review
  Interventions: Diagnostic Test: Pharmacogenomics testing; Other: Pharmacist review

INTERVENTIONS:
Diagnostic Test: Pharmacogenomics testing — Participants will undergo pharmacogenomics testing and will be asked to provide a one-time buccal scraping. These results will be utilized for clinical treatment decisions.
  Arms: Intervention Group B
Other: Pharmacist review — Participants will have their medical information, including patient demographics, problem list, medication list, allergies, and relevant lab work reviewed by a One Point pharmacist. The pharmacist will work with the Palliative Medicine team to make medication related recommendations to improve individual patient care. The pharmacist will call the patient roughly 48 hours following their outpatient consultation or hospital discharge to review the medication list and address any medication-related questions. The pharmacy will send refill reminders to the patients.
  Arms: Intervention Group A; Intervention Group B

SUMMARY:
Researchers are trying to learn more about how pharmacists and pharmacogenomic testing can help care providers improve control of symptoms and quality of life in seriously ill patients.

DETAILED DESCRIPTION:
Participants in the study will be randomized to A) standard of care, B) standard of care with medication therapy management provided by a pharmacist, or C) standard of care with medication therapy management by a pharmacist who has access to the patient's pharmacogenomics profile accessible to guide them. We will be measuring level of symptom control in each group over the subsequent 6 months.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age 18 years and older
* Palliative Medicine is consulted for the first time in either the outpatient setting for symptom management and plan to continue to follow up with the Palliative Medicine team in the outpatient setting for the foreseeable future.
* Insurance accepted at Mayo Clinic Arizona.
* Live within metro Phoenix area.

Exclusion Criteria:

* Vulnerable adults
* Under 18 years of age
* Pregnant Patients
* Subjects whose medical insurance requires use of specific pharmacies
* Non English Speaking Patients
* Patients that lack capacity for medical decision making
* Patients who live outside the metro Phoenix area
* Patients who are lost to follow up secondary to enrolling in hospice, die or failure to show or answer surveys within 2 months of enrollment.
* Patient with uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent.
* Patient's previously established within the Palliative Medicine Clinic who receive ongoing Palliative Medicine services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Change in symptom control | Baseline,1, 2, 4, and 6 months
  Measure using the self-reported Edmonton Symptom Assessment scale where a lower score indicates good symptom control and higher score indicates poor symptom control

CONTACTS AND LOCATIONS:
Overall Officials: Mark Edwin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials